CLINICAL TRIAL: NCT05732987
Title: Case-Control Study of the Genetic Architecture of Neutrophil-Mediated Inflammatory Skin Diseases
Brief Title: Genetic Architecture of Neutrophil-Mediated Inflammatory Skin Diseases
Acronym: NEUTROSKIN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02645; sp19Navarini3
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Neutrophil-mediated Inflammatory Dermatoses; Inflammatory Dermatoses
Keywords: inflammasome; inflammation-driving pathway; gene variants; next generation sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All samples originating from biobanks or Dermatology USB (fixed tissue) will be returned to origin after finishing of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Biobank- samples from NMID patients: 600 samples from NMID patients from the Biobank Dermatology Unispital Basel (USB) (Biobank USB) and from the biobank of the Dermatology Department of the University Hospital Zürich (USZ) (Biobank USZ) will be included.
  Interventions: Other: Analysis of samples
- Formalin-fixed and paraffin-embedded (FFPE) samples: About 50 of formalin-fixed and paraffin-embedded (FFPE) samples from the Dermatology USB collected before 2014 for RNA and protein expression analyses will be reused. The patients in questions are informed about the study and the coded use of their samples.
  Interventions: Other: Analysis of samples
- Biobank- samples from controls: 2'700 anonymized control genomes as well as 150 anonymized control samples for the proteomics approach can be used as control samples from the biobank of the Dermatology Department of the University Hospital Zürich (Biobank Dermatology USZ).
  Interventions: Other: Analysis of samples
- Fresh skin samples from healthy donors: A maximum of 20 fresh skin samples from healthy donors are required per skin location. They will be requested from healthy volunteers after information about the study and receiving the informed consent.
  Interventions: Other: Analysis of samples

INTERVENTIONS:
Other: Analysis of samples — DNA extraction from blood or saliva samples for the identification of gene variants by next generation sequencing;
Other: Analysis of samples — RNA extraction from blood and skin samples for Nanostring analyses, quantitative RT-PCR or RNA sequencing.
Other: Analysis of samples — Biobanked skin samples will be analyzed by immunostaining and imaging techniques to identify cell types in lesions and compare them to healthy skin.
Other: Analysis of samples — Cells isolated from biobanked blood and skin samples will be cultured in vitro and proteins will be analyzed by ELISA (secreted proteins) and western blot (cell proteins).

SUMMARY:
This study is to identify rare, disease-causing mutations of several rare neutrophil dermatoses. To identify associations between NMID and variants in the genome next generation sequencing, mainly whole exome sequencing, will be used. In a second approach the expression level of already known inflammatory proteins in skin samples will be investigated.

DETAILED DESCRIPTION:
The origin of rare severe inflammatory skin diseases in dermatology is insufficiently known. They have in common the presence and activation of phagocytes, affect the quality of life through pain and inflammation and disfiguration, and can even be fatal. This study is intended to build on the findings that several of these neutrophil-mediated inflammatory dermatoses (NMID) have a genetic background and to identify rare, disease-causing mutations of several rare neutrophil dermatoses. This non-clinical case-control study is a research project with biological material and health-related data. To identify associations between NMID and variants in the genome next generation sequencing, mainly whole exome sequencing, will be used. In a second approach the expression level of already known inflammatory proteins in skin samples will be investigated. The data are obtained and verified using standardized methods as e.g. Nanostring, RNA sequencing and qRT-polymerase chain reaction (PCR), proteomics assays and immunohistochemistry as well as flow cytometry and imaging mass cytometry, ELISA, and Western Blot.

ELIGIBILITY:
Inclusion Criteria:

* written consent of the participating person
* diagnosis of a disease in the NMID form group or proband of the control group

Exclusion Criteria for patients:

* Missing informed consent if samples collected after 2014
* no diagnosis of NMID

Exclusion Criteria for healthy controls:

* Missing informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants will largely be recruited by a.) prospectively collected biopsies of patients from biobanks or b.) analyzing, contacting, and including/excluding the existing patient population of our clinic (FFPE tissues).
  Healthy skin is obtained from patients undergoing plastic surgery at the USB. These patients will be informed and their informed consent obtained before surgery.
Sampling Method: Probability Sample
Enrollment: 3370 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Number of protein-coding rare variants associated with forms of NMID | one time assessment at baseline
  The primary endpoint consists in the determination of association between newly identified or previously reported rare gene variants and one or more forms of NMIDs. The discovery of such genetic variants will lead to the identification of defective molecular mechanisms involved in abnormal cutaneous immune reactions in these patients: - Statistically significant association between genetic data and NMID
  * Detection of protein-coding rare variants associated with forms of NMID
  * Identification of inflammasome activation in different stages of NMID

SECONDARY OUTCOMES:
Imaging Mass Cytometry | one time assessment at baseline
  The secondary endpoint will consist in the determination of consequences at the molecular and cellular levels of gene variants and subsequently encoded proteins in the cutaneous lesions from NMID patients by the measurement of protein interactions and networks, immune cells, cytokines and receptors in forms of NMID by statistically significant association of selected reaction monitoring results including: -Imaging Mass Cytometry
RNA expression | one time assessment at baseline
  The secondary endpoint will consist in the determination of consequences at the molecular and cellular levels of gene variants and subsequently encoded proteins in the cutaneous lesions from NMID patients by the measurement of protein interactions and networks, immune cells, cytokines and receptors in forms of NMID by statistically significant association of selected reaction monitoring results including: - RNA expression
Immune cell count | one time assessment at baseline
  The secondary endpoint will consist in the determination of consequences at the molecular and cellular levels of gene variants and subsequently encoded proteins in the cutaneous lesions from NMID patients by the measurement of protein interactions and networks, immune cells, cytokines and receptors in forms of NMID by statistically significant association of selected reaction monitoring results including: - Immune cell count
Rate of mean fluorescence intensity of immune cells | one time assessment at baseline
  The secondary endpoint will consist in the determination of consequences at the molecular and cellular levels of gene variants and subsequently encoded proteins in the cutaneous lesions from NMID patients by the measurement of protein interactions and networks, immune cells, cytokines and receptors in forms of NMID by statistically significant association of selected reaction monitoring results including: - Mean fluorescence intensity of immune cells
Protein quantification (ELISA) | one time assessment at baseline
  The secondary endpoint will consist in the determination of consequences at the molecular and cellular levels of gene variants and subsequently encoded proteins in the cutaneous lesions from NMID patients by the measurement of protein interactions and networks, immune cells, cytokines and receptors in forms of NMID by statistically significant association of selected reaction monitoring results including: - Protein quantification (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Navarini, Prof. Dr. med., Principal Investigator — University Hospital Basel, Clinic of Dermatology
Locations (1):
- University Hospital Basel, Clinic of Dermatology, Basel, Switzerland